CLINICAL TRIAL: NCT01839214
Title: A Randomized, Double-Blind, 12-Week, Placebo-Controlled Study Followed by a 12-Week Extension Phase Without Placebo to Evaluate the Efficacy and Safety of Oral VB-201 in Subjects With Mild to Moderate Ulcerative Colitis
Brief Title: A Study to Evaluate the Efficacy and Safety of VB-201 in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VB-201-064
Record Dates: First submitted 2013-04-21; First posted 2013-04-24 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — 1-palmityl-2-(4-carboxybutyl)-sn-glycero-3-phosphocholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VB-201 160mg (Experimental): Subjects will received 80mg twice daily for 24 weeks.
  Interventions: Drug: VB-201 160mg
- Placebo with crossover to VB-201 160mg (Placebo Comparator): Subjects on placebo will crossover to VB-201 160 at week 12.
  Interventions: Drug: VB-201 160mg; Drug: Placebo

INTERVENTIONS:
Drug: VB-201 160mg
Drug: Placebo
  Arms: Placebo with crossover to VB-201 160mg

SUMMARY:
This study will examine the safety and efficacy in subjects with mild to moderate ulcerative colitis, as measured by Modified Mayo Score, Modified Baron Score, IBDQ, calprotectin and other assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 years of age, who has a diagnosis of active UC for at least 6 months prior to screening
* A rectal/colonic biopsy obtained previously and consistent with a diagnosis of UC
* Endoscopy (flexible sigmoidoscopy unless surveillance colonoscopy is clinically indicated) confirming diagnosis of UC within 2 weeks prior to randomization
* Endoscopy (flexible sigmoidoscopy unless surveillance colonoscopy is clinically indicated) confirming diagnosis of UC within 2 weeks prior to randomization
* Active UC despite previous treatment with at least one 5-ASA compound at a dose of ≥2000 mg/day for at least 4 weeks or documented intolerance to such therapy

Exclusion Criteria:

* Diagnosis of indeterminate colitis, Crohn's disease, or clinical findings suggestive of Crohn's disease (fistula or granulomas on biopsy) or microscopic colitis (collagenous colitis or lymphocytic colitis)
* Subject whose symptoms are likely caused by factors other than inflammatory UC, including infection or irritable bowel syndrome (IBS)
* History of dysplasia on colonic biopsy
* Subject with ≥ 8 year history of pancolitis or ≥ 15 year history of left sided colitis unless a colonoscopy with surveillance biopsies to screen for colon cancer has been performed within the past year
* Subject ≥ 50 years of age who has not had a colonoscopy to screen for colorectal polyps and colon cancer within the past 5 years
* Subject who has had any prior surgical resection of any part of the colon excluding the appendix
* Previous treatment with any biologic product including investigational biologic products within 1 year prior to baseline visit
* The subject is taking Systemic corticosteroids, Azathioprine/6-mercaptopurine/methotrexate, immunosuppressants, Oral 5-ASA compounds unless they have been on a stable dose of sufficient duration prior to Baseline. If recently discontinued the subject must have had a wash-out periods of sufficient duration prior to Baseline
* Rectally administered corticosteroids or 5-ASA, antibiotics for the treatment of UC and probiotics within 14 days of the Baseline Visit and throughout the study
* The subject has with a stool culture positive for pathogenic ova or parasites, enteric pathogens or Clostridium difficile toxin at the Screening Visit
* Presence of, or history of cancer, with the exception of skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Modified Mayo Score indicating remission | Week 12 and Week 24
  The proportion of subjects in remission at Weeks 12 and 24 in the VB-201 160mg (80 mg BID) treatment group compared to placebo group.

SECONDARY OUTCOMES:
Modified Mayo Score indicating response | Week 12 and Week 24
  The proportion of subjects responding at Weeks 12 and 24 in the VB-201 160mg (80 mg BID) treatment group compared to placebo group.

OTHER OUTCOMES:
Frequency of Adverse Events | From Baseline through safety follow up at Week 28
  As measured by changes from baseline in physical exam, vital signs, ECG, concomitant medications, laboratory values.
Reduction in Modified Mayo Score | Week 12 and Week 24
  The proportion of subjects in each arm with a 2-point or greater decrease in the Modified Mayo score at Weeks 12 and 24.
Modified Baron Score | Week 12 and Week 24
  Change in the modified Baron score from Baseline to Weeks 12 and 24 in the VB-201 treatment group as compared to the placebo group.
Mucosal Healing | Wee 12 and Week 24
  The proportion of subjects in each arm with mucosal healing at Weeks 12 and 24 in the VB-201 treatment group compared to placebo group.

CONTACTS AND LOCATIONS:
Locations (3):
- VBL Investigative Site, Sofia, Bulgaria
- VBL Investigative Site, Szombathely, Hungary
- VBL Investigative Site, Warsaw, Poland